CLINICAL TRIAL: NCT00563186
Title: Physical Plant Design and Engineering Controls and the Prevention of Nosocomial Infections and Antibiotic Resistant Organism Colonization Events - A Proposal for a Prospective Controlled Trial
Brief Title: Hospital Design and Risk of Nosocomial Infections: A Prospective Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Calgary Health Region (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Alberta Heritage Foundation for Medical Research (Other)
Responsible Party: Principal Investigator, Dr. John Conly, Dr John Conly, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CIHR-PHE-81963
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Results first posted 2018-10-23 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Vancomycin Resistant Enterococci Infection; Clostridium Difficile Infection; Nosocomial Infection; Methicillin Resistant Staphylococcus Aureus Infection (MRSA)
Keywords: infection control; nosocomial infection; hospital design; physical plant design; antibiotic resistant organisms; MRSA; VRE; CDI
MeSH Terms: conditions — Clostridium Infections; Cross Infection

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Experimental): Admission to a novel hospital ward (e.g. abundance of sinks, predominance (80%) of private rooms, absence of shared bathrooms, absence of curtains)
  Interventions: Other: Admission to a novel hospital ward
- B (No Intervention): Hospital admission to a ward with traditional design features (eg. lack of sinks, predominance of 4-bed rooms [80%], shared bathrooms, curtains present)

INTERVENTIONS:
Other: Admission to a novel hospital ward — Hospital admission to a ward with novel infection control design features (e.g., abundance of sinks, predominance (80%) of private rooms, absence of shared bathrooms, absence of curtains)
  Arms: A

SUMMARY:
With the construction of a new medical teaching ward with features designed to reduce hospital-acquired infections, we hypothesized that the design of the new ward was the major factor that contributed to the improved outcomes and designed a prospective, controlled study to examine this hypothesis.

DETAILED DESCRIPTION:
Recent studies have underscored the importance of optimizing design standards to maximize patient and health care worker safety, including the prevention of hospital acquired infections (HAI) in patients. Health care associated infections are a major contributor to adverse events in healthcare, estimated to occur in 3-20% of all acute care admissions in Canada. A review of the role of the physical environment and adverse events identified no prospective randomized controlled trials of physical plant design and its impact on hospital acquired infections. With the construction in 2004 of a unique $5-million, 36-bed medical teaching unit at Foothills Medical Centre (FMC) with a prototypical design with features to reduce HAI and an overarching mandate to test new concepts in health care delivery, the opportunity exists to rigorously study the impact of design, construction and engineering controls (DCECs) on specific hospital acquired infections and antibiotic resistant organism (ARO) colonization. In the first year of operation the incidence density of hospital acquired infections and/or colonization with marker organisms has declined by almost 70%. Given that there were no changes in the types of patients, medical, nursing or housekeeping staff, we hypothesized that the design of the new ward was the major factor which contributed to the improved outcomes. Given the pre-post study design we are uncertain as to which factor is most important in reducing HAI /colonization rates.

We therefore propose to conduct a prospective, controlled investigator blinded trial of the impact of DCECs on specific HAIs and ARO colonization. We propose to allocate general medical patients, with an allocation scheme that incorporates randomness, to one of 2 types of medical wards at the FMC, either "historic design" wards (ie control wards in the non-renovated portions of FMC or Unit 36 (the experimental new design ward). The medical wards are very similar with respect to the patient mix, acuity of care, medical staff, nursing staff and skill mix, educational levels, housekeeping and levels of knowledge about infection control practices but differ in design. Variables which may otherwise have confounded the outcome of hospital acquired infections/colonizations may be controlled allowing the effect of the differences in design, construction and engineering controls to be studied. The older design wards have predominantly 4-bed and some 2-bed rooms with shared bathrooms, less space and fewer handwashing sinks/patient. The study will require 9750 patient days of observation in the "historic design"wards and 19,500 patient days of observation in Unit 36 to ensure 80% statistical power to detect a 60% difference in the rates of incident cases of selected HAIs and ARO colonizations (the primary outcome measure) with an α level of 0.05 assuming that incident cases in each unit follow Poisson distribution based on well established historic trends on these units.

In addition we propose to add a nested mixed methods social science study within the construct of the prospective study to understand the fit between the health care workers and the physical environment. In recognition that the proposed intervention may be defined as a "complex intervention" with HAIs affected by many factors related to physical plant design, organizational factors, and health care worker practices, it was considered prudent to measure and describe worker and organizational factors on the medical inpatient care units included in the proposed intervention.

Our proposed study is being done with the collaboration and support of both the Operations and Planning & Capital Development portfolios of the Calgary Health Region. The Region is in the throes of a major expansion with over $1 billion of new capital health care developments and the addition of over 700 new beds by 2010. The finding of favorable outcomes on the medical ward with its special design, construction and engineered controls in a well designed prospective study of this nature would be the first of its kind and has the potential to change the fundamental design of new medical wards in the Calgary Health Region and in other jurisdictions within Canada.

ELIGIBILITY:
Inclusion Criteria:

* are adults aged 18 or older with medical diagnoses being admitted to one of three in-hospital general medical services at the FMC (one of the two in-patient General Internal Medicine services at the FMC)
* are admitted via the emergency room
* are admitted from the urgent assessment clinic or the community

Exclusion Criteria:

* are admitted from another acute care medical institution
* require telemetry monitoring of their cardiac rhythm (a specific medical situation that dictates need for admission to a nonUnit 36 bed).
* have other clinical circumstances (eg clinical instability) mandating a physician to indicate clinical preference for admission of the patient to a specific location in the hospital
* are admitted from the intensive care unit or another hospital ward
* are admitted for less than 48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1514 (Actual)
Dates: Start 2007-06; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John M Conly, MD, Principal Investigator — University of Calgary; William A Ghali, MD, Principal Investigator — University of Calgary; Manuel Mah, MD, Principal Investigator — Calgary Health Region; Donna Holton, MD, Principal Investigator — Calgary Health Region; Elizabeth A Henderson, PhD, Principal Investigator — University of Calgary; Peter Faris, PhD, Principal Investigator — University of Calgary; Jean Wallace, PhD, Principal Investigator — University of Calgary
Locations (1):
- Foothills Hospital, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
Published: J Ellison, D Southern, D Holton, et al. Hospital ward design and prevention of hospital-acquired infections: A prospective clinical trial. Can J Infect Dis Med Microbiol 2014;25(5):265-270.
  Data was coded and entered into a computer for analysis and was non-nominal to protect the privacy of the information. Since the data were bed-specific, we will not be sharing the de-identified data.

REFERENCES:
- See also: Website for the Medical Ward of the 21st Century Initiative. — http://www.w21c.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between June 2007 and February 2010 all patients admitted to the General Internal Medicine Service at Foothills Medical Centre from the emergency room, urgent assessment clinic or the community were assessed for eligibility into the study.
Pre-assignment Details: Exclusions: admitted from another health care facility or another hospital ward or to a non-study unit, required telemetry, < 18 years of age, or were preferentially admitted to the novel or the traditional design ward. Once pre-assigned, excluded if LOS <48 hours (Novel ward=97, Historic ward=74); or data incomplete (Novel ward=1; Historic ward=1)
Groups:
- Novel Hospital Ward Admission: Hospital admission to a ward with novel infection control design features (e.g. abundance of sinks, predominance (80%) of private rooms, absence of shared bathrooms)
- Traditional Hospital Ward Admission: Hospital admission to a ward with traditional infection control design features (e.g. lack of sinks, predominance (80%) of 4-bed rooms, shared bathrooms)
Period: Overall Study
Arm/Group | Novel Hospital Ward Admission | Traditional Hospital Ward Admission
Started | 1008 (Patients allocated to the Novel Hospital Ward) | 679 (Patients allocated to the Traditional Hospital Ward)
Completed (excluded if length of stay (LOS)<48 hours or incomplete data) | 910 | 604
Not Completed | 98 | 75
Not completed — LOS<48 hours | 97 | 74
Not completed — Incomplete data | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Novel Hospital Ward Admission | Traditional Hospital Ward Admission | Total
Number analyzed (Participants) | 910 | 604 | 1514
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 400 | 305 | 705
  >=65 years | 510 | 299 | 809
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.62 (18.44) | 63.22 (18.78) | 61.66 (18.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 407 | 278 | 685
  Male | 503 | 326 | 829
Region of Enrollment [Number; unit: participants]
  Canada | 910 | 604 | 1514

OUTCOME MEASURES:

1. Primary Outcome: Incidence Density of Hospital-acquired Infection With Clostridium Difficile (CDI), and Hospital-acquired Infection or Colonization With Vancomycin-resistant Enterococcus (VRE), or Methicillin-resistant Staphylococcus Aureus (MRSA).
Time Frame: participants were followed for the duration of hospital stay, an average of 10 days
Population: All patients meeting inclusion criteria, and admitted to the General Internal Medicine (GIM) service on the novel infection control design ward or the traditional infection control design ward were followed for the development of MRSA or VRE infection (inf) or colonization (col) or CDI after 48 hours of admission
Measure: Number; unit: events per 1000 patient days
Arm/Group | Novel Hospital Ward Admission | Traditional Hospital Ward Admission
Number analyzed (Participants) | 910 | 604
events per 1000 patient days
  CDI | 1.16 | 0.84
  MRSA Infections / Colonizations | 1.27 | 1.01
  VRE Infections / Colonizations | 0.53 | 0
  Overall Total Infections / Colonizations | 2.96 | 1.85
Statistical Analysis 1: Comparison: Novel Hospital Ward Admission vs Traditional Hospital Ward Admission; It was calculated that this study will require 9750 patient days of observation in the "traditional design" wards and 19,500 patient days of observation in the "novel design" ward to ensure 80% statistical power to detect a 60% difference in the rates of incident cases of selected HAIs and ARO colonizations (the primary outcome measure) with an α level of 0.05 assuming that incident cases in each unit follow Poisson distribution based on well established historic trends on these units; Test type: Superiority or Other — This statistical analysis applies to the overall VRE, CDI and MRSA infection and colonization events expressed as incidence density (per 1000 patient-days at risk); p = 0.18, Poisson; Incidence Rate ratio = 1.60, 95% CI 2-sided [0.80 to 3.22], Standard Error of Mean 0.57 — Numerator is novel ward and denominator is traditional ward

2. Secondary Outcome: Number of MRSA, VRE and CDI Occurring in Single-bed Rooms vs. Multiple Bed Rooms AND Occurring in Outbreaks Related to the Primary Case
Description: If a patient is swabbed and found to be positive (for MRSA or VRE), their current roommate\roommates will be swabbed (if in the same room > 48 hrs) as well as any other patient that shared a room with this patient for > 48 hours during this stay. Any patient who may have shared a bathroom with the first patient would also be swabbed. If the results from this investigation showed any positive roommates, then the process would repeat for each positive patient. Then, in consult with the infectious disease physician, a call will be made regarding a point prevalence study to determine the attack rate\burden of disease on the unit.
Time Frame: in-hospital
Population: An outbreak occurred when more than 1 case of MRSA, VRE or CDI was epidemiologically linked to a primary case. In total 22 outbreak cases were detected during the study. The location of these outbreak cases (single-bed rooms vs. multi-bed rooms) was identified in the Novel Hospital Ward and the Traditional Hospital Ward
Measure: Number; unit: outbeak infections/colonizations
Units Other Than Participants: Total Number of Outbreak cases
Groups:
- Novel and Traditional Hospital Ward Admission: Number of MRSA, VRE and CDI cases occurring in single-and multiple-bed rooms in Novel Hospital Ward and Traditional Hospital Ward during outbreaks
Arm/Group | Novel and Traditional Hospital Ward Admission
Number analyzed (Participants) | 1514
Number analyzed (Total Number of Outbreak cases) | 22
outbeak infections/colonizations
  Single-bed Rooms | 3
  Multiple-bed rooms | 19

3. Post Hoc Outcome: Event Incidence Density in Single vs Multi-bed Rooms in Novel Design Ward Only
Description: The incidence density of MRSA, VRE and CDI occurring in single-bed vs. multi-bed rooms was examined on only the novel design ward
Time Frame: In-hospital
Population: All patients that met the inclusion and exclusion categories and were admitted to the novel design ward were assessed for the development of MRSA, VRE or CDI. The incidence densities in single-bed rooms were then compared to the incidence densities in multiple-bed rooms.
Measure: Number; unit: events per 1000 patient days
Groups:
- Incidence Density in Single-bed Rooms: # MRSA, VRE and CDI (expressed per 1000 pt days)occurring in single-bed rooms on the novel design ward
- Incidence Density in Multi-bed Rooms: # MRSA, VRE and CDI (expressed per 1000 pt days)occurring in multi-bed rooms on the novel design ward
Arm/Group | Incidence Density in Single-bed Rooms | Incidence Density in Multi-bed Rooms
Number analyzed (Participants) | 256 | 654
events per 1000 patient days | 1.89 | 3.47
Statistical Analysis 1: Comparison: Incidence Density in Single-bed Rooms vs Incidence Density in Multi-bed Rooms; Test type: Superiority or Other; p = 0.175, Large test for person-time analysis; Rate Ratio = 1.929, 95% CI 2-sided [0.76 to 4.9], Standard Error of Mean 0.493

ADVERSE EVENTS:
Arm/Group | Novel Hospital Ward Admission | Traditional Hospital Ward Admission
Serious Adverse Events (participants affected / at risk) | 0/910 | 0/604
Other Adverse Events (participants affected / at risk) | 0/910 | 0/604

LIMITATIONS AND CAVEATS:
Chronic overcapacity issues impacted the ability to truly randomize which may have introduced a selection bias,there was an unanticipated conversion of single rooms to multi-bed rooms on the novel ward, limited generalizability outside GIM patients

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes